CLINICAL TRIAL: NCT04498221
Title: Prospective, Multi-Centre, Phase II Validation Study for a Lymphatic Imaging Protocol in Establishing Drainage Patterns in Patients With Oropharyngeal Cancer
Brief Title: Lymphatic Mapping Of Oropharyngeal Cancer
Acronym: LOOC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University College, London (Other)
Collaborators: National Institute for Health Research, United Kingdom (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 127659
Record Dates: First submitted 2019-12-04; First posted 2020-08-04 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Oropharyngeal Cancer
MeSH Terms: conditions — Oropharyngeal Neoplasms | interventions — X-Rays; Surgical Procedures, Operative

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Imaging Phase (Experimental): During routine examination under anaesthetic 4 x peritumoural injection of investigator's choice of 99mTc-human albumin colloidal particles or Lymphoseek (lymphatic mapping tracer) followed by freehand SPECT scan
  Interventions: Procedure: Imaging procedure
- Surgical Phase (Experimental): Excision of contralateral nodes identified on imaging *(fhSPECT or SPECT/CT*) during routine examination under anaesthetic. Serial sectioning of excised (sentinel) nodes to identify micrometastasis.
  Interventions: Procedure: Surgical procedure

INTERVENTIONS:
Procedure: Imaging procedure — During routine examination under anaesthetic 4 x peritumoural injection of investigator's choice of 99mTc-human albumin colloidal particles or Lymphoseek (lymphatic mapping tracer) followed by freehand SPECT scan
  Arms: Imaging Phase
Procedure: Surgical procedure — Excision of contralateral nodes identified on imaging *(fhSPECT or SPECT/CT*) during routine examination under anaesthetic. Serial sectioning of excised (sentinel) nodes to identify micrometastasis.
  Arms: Surgical Phase

SUMMARY:
A multi-centre validation study to evaluate whether a new imaging and surgical protocol would work as well as the current gold standard in identifying sentinel nodes in patients with oropharyngeal cancer.

DETAILED DESCRIPTION:
Cancer at the back of the mouth and throat is usually discovered after it has spread to lymph glands in the neck. Treatment therefore involves dealing with both the original tumour (in the mouth/throat) and the spread cancer in the lymph glands. This type of cancer sometimes spreads to both sides of the neck, not just the side on which the original tumour was located. The decision as to whether to treat the other side of the neck as well depends on various factors including the aggressiveness of the tumour, whether the patient smokes and whether or not the Human Papilloma Virus (HPV) is present in the tumour. This is inevitably inexact, and assessing the likelihood of the cancer spreading to the other side of the neck always involves an element of estimation. Some patients end up being treated unnecessarily on both sides (often with severe and lasting effects on swallowing, meaning they have to use a feeding tube), while others receive treatment on one side only but the cancer comes back on the other side.

This study will provide more accurate information on which to base the decision as to whether to treat the other side of the neck. The study will use a procedure known as sentinel node biopsy (SNB) to establish (with a high degree of accuracy) whether or not the cancer has spread to the other side of the neck. The study will be in two stages. The first stage is the imaging stage. A very low does of a radioactive tracer substance will be injected into the tumour. The radioactive tracers used in this study are either Human albumin colloidal particles or Lymphoseek. Once injected, they move quickly into the lymph nodes and can then be detected using a handheld gamma camera. The first nodes that the radiotracer moves into are the "sentinel" nodes. Patients already undergo an examination under anaesthetic (EUA); the patients participating in the study will have the radiotracer injected additionally and the sentinel nodes detected during this EUA. The use of the handheld camera is relatively new; so, all of the patients in the study will also have a CT scan the next day to double check whether the handheld camera identified the sentinel nodes correctly. The second stage of the study, the surgery stage, will involve a new group of patients having the imaging procedure. Those who do have sentinel nodes in the other side of the neck will have them removed during the EUA. Those nodes will then be examined thoroughly for signs of cancer. A separate limb of stage one of the study will involve some patients whose main tumours are easily accessible also having their tumour injected with the radiotracer a second time under local anaesthetic in an outpatient clinic. In the study this will take place several days after the initial injection with the radiotracer. If this procedure is found to be acceptable to patients, it would mean that patients could have the radiotracer injected before the EUA, thereby allowing time for the sentinel nodes to be identified by CT scan so that they can be removed during the EUA. This will provide a way to ensure that, even if the handheld camera cannot be used, the sentinel nodes can still be removed while the patient is under anaesthetic for the EUA. If the study is successful, the patient will be able to have much more accurate information about whether their cancer has, or might, spread to the other side of the neck, without having to undergo an additional general anaesthetic.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 or over
* New diagnosis of OPC - all anatomical subsites and HPV status accepted
* Unilateral metastatic nodes equating to AJCC TNM8 clinical staging N1-N2b for P16 negative and N1 for P16 positive patients.

Exclusion Criteria:

* Suspicious bilateral nodes on imaging
* Previous radiotherapy or surgery to the neck
* Second primary oropharyngeal tumours
* Distant metastasis (e.g. lung, bone)
* Pregnancy and lactation
* Inability to give informed consent
* Allergy to lymphatic tracers

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2022-07-07 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Rate of contralateral drainage | 24 hours post injection
  Rate of contralateral drainage
Accuracy of detection of contralateral nodes by lymphoscintigraphy using fhSPECT compared to SPECT/CT | 24 hours post injection
  Accuracy of detection of contralateral nodes by lymphoscintigraphy using fhSPECT compared to SPECT/CT
Number of contralateral nodes on SPECT/CT | 24 hours post injection
  Number of contralateral nodes on SPECT/CT will be used as the denominator in calculating the sensitivity of fhSPECT in independently verified images
Number and location of contralateral nodes seen with lymphoscintigraphy performed by i) single injection ii) four peritumoural injections (standard practice) as assessed by paired SPECT/CT scans. | 24 hours post injection
  Number and location of contralateral nodes seen with lymphoscintigraphy performed by i) single injection ii) four peritumoural injections (standard practice) as assessed by paired SPECT/CT scans.
Acceptability to patients assessed by questionnaire. | 24 hours post injection
  Acceptability to patients assessed by questionnaire.
Occult metastasis rate of contralateral nodes (positive sentinel node biopsy). | 24 hours post injection
  Occult metastasis rate of contralateral nodes (positive sentinel node biopsy).

CONTACTS AND LOCATIONS:
Overall Officials: Clare Schilling, Principal Investigator — University College, London
Locations (2):
- United Kingdom (2):
  - St George's University Hospitals NHS Foundation Trust, London
  - University College Hospital, London

IPD SHARING:
Plan to Share IPD: No
No identifiable data will be shared with anyone outside the study

REFERENCES:
- [Derived] Schilling C, Payne K, Wan S, Brew-Graves C, Ofo E, Ambler G, Weller A, Gnanasegaran G, Paleri V, Shaw R, Fleming J, Walker D, Bajwa M, McGurk M. Lymphatic mapping Of Oropharyngeal Cancer (LOOC): protocol for a phase II surgical imaging trial to evaluate contralateral drainage and occult metastasis in oropharyngeal cancer. BMJ Open. 2025 Jun 5;15(6):e101746. doi: 10.1136/bmjopen-2025-101746. PMID 40473291